CLINICAL TRIAL: NCT01730807
Title: IntellaTip MiFi XP Ablation Catheters First in Human Use Trial
Brief Title: IntellaTip MiFi XP Ablation Catheter Trial
Acronym: MiFi-CTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiFi-CTI
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Atrial Flutter
Keywords: Atrial Flutter; Ablation; Type I Atrial Flutter; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IntellaTip XP MiFi (Experimental): Patients with Atrial Flutter will receive ablation treatment with the IntellaTip MiFi XP catheter
  Interventions: Device: IntellaTip MiFi XP Catheter

INTERVENTIONS:
Device: IntellaTip MiFi XP Catheter — Temperature controlled ablation catheter

SUMMARY:
A study to assess the performance of a new catheter design for the treatment of Atrial Flutter.

DETAILED DESCRIPTION:
A prospective, non-blinded, single arm, single center study designed to assess the performance of the IntellaTip MiFi XP Ablation Catheter for the treatment of recurrent or sustained type I atrial Flutter.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* indicated for ablation for Atrial Flutter

Exclusion Criteria:

* Thrombus
* Recent MI/cardiac revascularization
* Prosthetic Valves
* recent ablation for atrial flutter
* atrial flutter with reversible cause
* Class IV HF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Acute Procedural Success | one day
  The Demonstration of bi-directional isthmus block at the end of the ablation procedure

SECONDARY OUTCOMES:
Complication Rate at procedure | 7 days
  Determine major complications in patients exposed to the device, which occur within 7 days of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Prashanthan Sanders, MD, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia